CLINICAL TRIAL: NCT02306928
Title: Population Pharmacokinetics of Piperacillin in the Early Phase of Septic Shock - Does Standard Dosing Result in Therapeutic Plasma Concentrations?
Brief Title: PK Analysis of Piperacillin in Septic Shock Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristina Öbrink-Hansen, MD, University of Aarhus
Other Study IDs: PIP/TAZO-ICU
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Septic Shock
Keywords: Septic shock; Intensive care unit; Therapeutic drug monitoring; Pharmacokinetics; Critically ill
MeSH Terms: conditions — Shock, Septic; Critical Illness | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Piperacillin pharmacokinetics: Patients with suspected septic shock who are treated with piperacillin/tazobactam.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw

SUMMARY:
Antibiotic dosing in septic shock patients poses a challenge for clinicians due to the pharmacokinetic changes seen in this population. Piperacillin/tazobactam is often used for empirical treatment, and initial appropriate dosing is crucial for reducing mortality.

We determined the pharmacokinetic profile of piperacillin 4g every 8 hour in 15 patients treated empirically for septic shock. A PK population model was established with the dual purpose to assess current standard treatment and to simulate alternative dosing regimens and modes of administration. Time above the minimal inhibitory concentration (T>MIC) predicted for each patient were evaluated against clinical breakpoint MIC for Pseudomonas aeruginosa (16 mg/L). Pharmacokinetic-pharmacodynamic (PK-PD) targets evaluated were 100% f T>MIC and 50% fT>4xMIC.

DETAILED DESCRIPTION:
Early appropriate antimicrobial therapy is of utmost importance for reducing mortality in critically ill patients with sepsis and septic shock. Patophysiological changes associated with the septic process, such as changes in volume of distribution (Vd), drug clearance (CL), decrease in plasma-protein concentration and organ dysfunction, lead to pharmacokinetic (PK) changes that may alter the efficacy of the antimicrobial given. As a consequence, antibiotic plasma concentrations are variable and hard to predict in these patients, which makes optimal antibiotic exposure a challenge, especially in the early phase of treatment. In sepctic shock patients, appropriate dosing is even more important, as effective antimicrobial therapy within the first hour of documented hypotension is associated with increased survival to hospital discharge.

Piperacillin/tazobactam is a β-lactam - β-lactamase inhibitor combination frequently used for empirical treatment in the critically ill. It is a time-dependent antibiotic where antibacterial activity is related to the time for which the free, unbound concentation of the drug is maintained above the minimal inhibitory concentration (f T>MIC). Maximizing f T>MIC both increases the therapeutic impact and reduces the risk of drug resistance development. Because of the PK changes seen in the critically ill, standard dosing of antimicrobials may result in subtherapeutic plasma-concentrations (17) and it has been suggested that current empiric dosing recommendations for ICU patients are inadequate and needs to be reconsidered (18). Patients with septic shock are especially vulnerable (7) and optimal dosing in these patients is crucial for reducing mortality.

Piperacillin/tazobactam 4g/0.5g every 8 hour (h) is the empiric standard dosing for sepsis and septic shock. The aim of this study was to determine if this dosing results in therapeutic plasma concentrations in septic shock patients, within the initial 24 hours of therapy. A PK population model was established with the dual purpose to assess current standard treatment and to simulate alternative dosing regimens and modes of administration.

Critically ill patients with known or suspected septic shock who required noradrenaline infusion and who were prescribed piperaillin/tazobactam 4g/0.5g (Tazocin®) by the treating physician were eligible for the study. Patients on renal replacement therapy and patients under the age of 18 were not included.

Piperacillin/tazobactam 4g/0.5g was administered intravenously (i.v.) over 3 minutes every 8 h. Blood samples (4 mL) were collected by trained staff from an arterial catheter around the time of administration of the third consecutive infusion. Each patient had a total of eight blood samples drawn; before administration of the drug (time 0), at 10, 20, 30 minutes and 1, 2, 4 and 8 h after administration of the drug.

The unbound piperacillin plasma concentrations were determined using ultra high performance liquid chromatography. If a bacteria was isolated from a patient, a MIC to piperacillin was obtained using E-tests on Mueller-Hinton agar plates. These MICs as well as clinical MIC breakpoints according to the European Committee on Antimicrobial Susceptibility Testing (EUCAST) for Pseudomonas aeruginosa were used to evaluate the following PK/PD targets: 100% f T>MIC and 50% fT>4xMIC.

There was no intervention in the study.

ELIGIBILITY:
Inclusion Criteria:

Treatment with piperacillin/tazobactam for less than 24 hours. Treatment with noradrenaline. -

Exclusion Criteria:

Renal replacement therapy. Age under 18.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with known or suspected septic shock admitted to the ICU, treated with piperacillin/tazobactam.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Storgaard, MD, Study Director — Department of Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of anesthesiology and intensive care, Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Derived] Obrink-Hansen K, Juul RV, Storgaard M, Thomsen MK, Hardlei TF, Brock B, Kreilgaard M, Gjedsted J. Population pharmacokinetics of piperacillin in the early phase of septic shock: does standard dosing result in therapeutic plasma concentrations? Antimicrob Agents Chemother. 2015 Nov;59(11):7018-26. doi: 10.1128/AAC.01347-15. Epub 2015 Sep 8. PMID 26349823

RESULTS

PARTICIPANT FLOW:
Groups:
- Piperacillin Pharmacokinetics: Patients with known or suspected septic shock who who required noradrenaline infusion and who were prescribed piperaillin/tazobactam 4g/0.5g (Tazocin®) by the treating physician were eligible for the study. Patients on renal replacement therapy and patients under the age of 18 were not included.
  Included patients had plasma concentrations of piperacillin, being the active β-lactam component, determined. Age, gender, body weight, APACHE (Acute Physiology and Chronic Health Evaluation) score on admission, SOFA (Sequential Organ Failure Assessment) score on day of sampling, amount of noradrenalin-infusion given during the third dosing interval and presence of acute kidney failure (AKI) of each enrolled patient were registered.
Period: Overall Study
Arm/Group | Piperacillin Pharmacokinetics
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [59 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Body weight [Median (Inter-Quartile Range); unit: kg] | 80 [70.2 to 95]

OUTCOME MEASURES:

1. Primary Outcome: 100% f T>MIC: Free Piperacillin Concentration Maintained Above the MIC Throughout the Dosing Interval.
Description: The piperacillin plasma concentration-time profiles were best described by a two-compartment model. Each individual model predicted T>MIC was compared to clinical breakpoint MIC for P.aeruginosa (16 mg/L). The number of patients who achieved the pre-defined PK/PD target were reported.
Time Frame: Participants were followed up to the third dosing interval after initiation of piperacillin/tazobactam. An average of 24 hours.
Measure: Number; unit: participants
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 15
participants | 10

2. Secondary Outcome: The Maximum Concentration of Piperacillin (Cmax)
Description: Maximum plasma concentration was predicted for each individual based on the final model fit.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 15
mg/L | 546 [363 to 668]

3. Secondary Outcome: The Area Under the Plasma-concentration Time Curve Concentration-time Curve From 0-8 Hours After the Studied Dose (AUC 0-8)
Description: Area under the free plasma concentration-time curve (fAUC0-8) was predicted for each individual based on the final model fit.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg.hr/L
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 15
mg.hr/L | 1148 [739 to 2492]

4. Secondary Outcome: Trough Piperacillin Plasma Concentration (Cmin)
Description: Trough plasma concentration (Cmin) was predicted for each individual based on the final model fit.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 15
mg/L | 51.7 [10.7 to 159.4]

5. Primary Outcome: 50% fT>4xMIC: Free Piperacillin Concentration Maintained at a Level Fourfold the MIC for at Least 50% of the Dosing Interval.
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 15
participants | 12

ADVERSE EVENTS:
Groups:
- Piperacillin Pharmacokinetics: Serious and non-serious adverse advents were not collected.
Arm/Group | Piperacillin Pharmacokinetics
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes